CLINICAL TRIAL: NCT03655951
Title: Parent-Teen Communication to Resist Unhealthy Media Messages
Brief Title: Birds and Bees Research Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Innovation Research & Training (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: R44HD082968 (NIH)
Record Dates: First submitted 2018-08-13; First posted 2018-09-04 (Actual); Results first posted 2020-11-10 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-10

CONDITIONS: Sexual Behavior; Communication
MeSH Terms: conditions — Sexual Behavior; Communication

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Outcomes Assessor and Care Provider - NA This is a web-based study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resource 1 (Experimental): Web-based resource on adolescent sexual health
  Interventions: Behavioral: Web-based resource on adolescent sexual health
- Resource 2 (Active Comparator): Alternate web-based resource on adolescent sexual health
  Interventions: Behavioral: Alternate web-based resource on adolescent sexual health

INTERVENTIONS:
Behavioral: Web-based resource on adolescent sexual health — Web-based resource on adolescent sexual health than the intervention.
  Arms: Resource 1
Behavioral: Alternate web-based resource on adolescent sexual health — This is a different web-based resource on adolescent sexual health than the intervention.
  Arms: Resource 2

SUMMARY:
The goal of this efficacy study is to evaluate how different web-based resources affect parents' and children's sexual health knowledge; attitudes, efficacy, intentions, and behaviors about parent-adolescent communication; attitudes about media messages; and media message deconstruction skills. Parent consumer satisfaction with the resources will also be assessed.

DETAILED DESCRIPTION:
While the majority of the students will receive sexual education at least once between seventh and twelfth grade, the content that they will receive varies greatly. Thus, adolescents turn to other sources for information about sex including their parents and the media. However, many parents face challenges in being prepared to discuss sex with their adolescent child. While over eighty percent of parents are talking with their children ages 10-18 about issues related to sex, far fewer (60%) discuss more difficult sexual topics such as birth control. These findings suggest that there is a need for evidence-based resources that teach parents the skills needed to have effective conversations with their adolescent children about sexual health topics and media messages that promote early and risky sex.

ELIGIBILITY:
Inclusion Criteria:

* parent or legal guardian of a child in 7th, 8th, or 9th grade

Exclusion Criteria:

* not fluent in English
* does not have access to internet to complete study tasks

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 730 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2019-06-20 (Actual); Study Completion 2019-06-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- innovation Research & Training, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Resource 1 | Resource 2
Started (Randomized) | 358 | 372
Completed Pretest | 344 | 366
Completed (Completed posttest) | 319 | 351
Not Completed | 39 | 21
Not completed — Lost to Follow-up | 39 | 20
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Resource 1 | Resource 2 | Total
Number analyzed (Participants) | 358 | 372 | 730
Age, Categorical [Count of Participants; unit: Participants] — Population: 730 participants were randomized.710 completed pretest and 670 completed posttest.
  Participants
    number analyzed (Participants) | 344 | 366 | 710
    <=18 years | 172 | 183 | 355
    Between 18 and 65 years | 172 | 183 | 355
    >=65 years | 0 | 0 | 0
Sex/Gender, Customized [Number; unit: participants] — Population: 730 participants were randomized.710 completed pretest and 670 completed posttest. Participants could skip questions, so not all participants answered all questions.
  participants
    Female: number analyzed (Participants) | 344 | 366 | 710
    Female | 201 | 217 | 418
    Male: number analyzed (Participants) | 344 | 366 | 710
    Male | 129 | 139 | 268
    Non-binary or prefered not to disclose: number analyzed (Participants) | 344 | 366 | 710
    Non-binary or prefered not to disclose | 10 | 2 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: 730 participants were randomized. 710 completed pretest. 670 completed posttest. Participants could skip questions.
  Participants
    number analyzed (Participants) | 344 | 366 | 710
    Hispanic or Latino | 35 | 41 | 76
    Not Hispanic or Latino | 307 | 317 | 624
    Unknown or Not Reported | 2 | 8 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: 730 participants were randomized.710 completed pretest and 670 completed posttest. Participants could skip questions, so not all participants answered all questions.
  Participants
    number analyzed (Participants) | 344 | 366 | 710
    American Indian or Alaska Native | 2 | 2 | 4
    Asian | 5 | 6 | 11
    Native Hawaiian or Other Pacific Islander | 3 | 1 | 4
    Black or African American | 58 | 42 | 100
    White | 225 | 248 | 473
    More than one race | 39 | 49 | 88
    Unknown or Not Reported | 12 | 18 | 30
Region of Enrollment [Count of Participants; unit: Participants] — Population: 730 participants were randomized.710 completed pretest and 670 completed posttest. Participants could skip questions, so not all participants answered all questions.
  Participants
    United States: number analyzed (Participants) | 344 | 366 | 710
    United States | 344 | 366 | 710

OUTCOME MEASURES:

1. Primary Outcome: Change in Parent Reported Frequency of Parent-child Communication About Relationships, Sex, and Media From Pretest to Posttest
Description: Parent questionnaires ask participants how frequently they engage in parent-child communication about relationships, sex, and media. (1. Never; 2. Rarely; 3. Sometimes; 4. Often). Higher numbers represent a better outcome.
Time Frame: 1) pretest questionnaire; 2) posttest questionnaire - 4 weeks after pretest
Population: The number of participants analyzed for this measure differs from the numbers in the Participant Flow module due to the fact that not all participants completed questionnaires at all time points and participants were able to skip questions on the questionnaire.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Resource 1 | Resource 2
Number analyzed (Participants) | 137 | 150
score on a scale
  Pretest/baseline to Post test/Week 4 | 3.13 (.0688) | 3.03 (.0663)
  Pretest/baseline to Follow-up/24 weeks | 2.94 (.08) | 2.94 (.08)
Statistical Analysis 1: Comparison: Resource 1 vs Resource 2; Test type: Equivalence — To examine intervention effects, a residual difference score approach was used to provide an estimate of change from baseline and is assessed by regressing post-intervention scores onto baseline scores and the treatment variables; p = .20, Regression, Linear

2. Primary Outcome: Change in Child Reported Frequency of Parent-child Communication About Relationships, Sex, and Media From Pretest to Posttest
Description: Child questionnaires ask participants how frequently they engage in parent-child communication about relationships, sex, and media. (1. Never; 2. Rarely; 3. Sometimes; 4. Often). Higher numbers represent a better outcome.
Time Frame: 1) pretest questionnaire; 2) posttest questionnaire - 4 weeks after pretest
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Resource 1 | Resource 2
Number analyzed (Participants) | 123 | 136
score on a scale | 2.4 (.0827) | 2.44 (.0811)
Statistical Analysis 1: Comparison: Resource 1 vs Resource 2; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = .69, Regression, Linear

3. Primary Outcome: Change in Parent Reported Frequency of Parent-child Communication About Relationships, Sex, and Media From Pretest to Follow-up
Description: as for outcome 1
Time Frame: 1) pretest questionnaire; 3) follow-up questionnaire - 24 weeks after pretest
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Resource 1 | Resource 2
Number analyzed (Participants) | 144 | 139
score on a scale | 3.09 (.08) | 3.15 (.08)
Statistical Analysis 1: Comparison: Resource 1 vs Resource 2; Test type: Equivalence — To examine intervention effects, a residual difference score approach was used to provide an estimate of change from baseline and is assessed by regressing follow-up scores onto baseline scores and the treatment variables; p = .48, Regression, Linear

4. Primary Outcome: Change in Child Reported Frequency of Parent-child Communication About Relationships, Sex, and Media From Pretest to Follow-up.
Description: as for outcome 2
Time Frame: 1) pretest questionnaire; 2) follow-up questionnaire - 24 weeks after pretest
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Resource 1 | Resource 2
Number analyzed (Participants) | 131 | 138
score on a scale | 2.58 (.1) | 2.66 (.1)
Statistical Analysis 1: Comparison: Resource 1 vs Resource 2; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; p = .36, Regression, Linear

5. Secondary Outcome: Change in Parental Perceived Importance of Parent-child Communication About Relationship and Sexual Health From Pretest to Posttest
Description: Parent questionnaire asks participants to report on a 4-point scale (1 =not at all important - 4=very important) how important they think it is to engage in parent-child communication about several relationship and sexual health topics (e.g., reasons to wait to have sex). Item responses will be averaged, and higher values represent a better outcome.
Time Frame: 1) pretest questionnaire; 2) posttest questionnaire - 4 weeks after pretest
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Resource 1 | Resource 2
Number analyzed (Participants) | 142 | 150
score on a scale | 3.69 (.0217) | 3.71 (.0214)
Statistical Analysis 1: Comparison: Resource 1 vs Resource 2; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = .48, Regression, Linear

6. Secondary Outcome: Change in Parent Level of Comfort With Parent-child Communication About Relationship and Sexual Health From Pretest to Posttest
Description: Parent questionnaire asks participants to report on a 4-point scale (1=not at all comfortable - 4=very comfortable) how comfortable they are engaging in parent-child communication about several relationship and sexual health topics (e.g., reasons to wait to have sex). Item responses will be averaged, and higher values represent a better outcome.
Time Frame: 1) pretest questionnaire; 2) posttest questionnaire - 4 weeks after pretest
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Resource 1 | Resource 2
Number analyzed (Participants) | 140 | 151
score on a scale | 3.5 (.0359) | 3.44 (.0354)
Statistical Analysis 1: Comparison: Resource 1 vs Resource 2; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = .41, Regression, Linear

7. Secondary Outcome: Change in Parent Reservations About Parent-child Communication About Relationship and Sexual Health From Pretest to Posttest
Description: Parent questionnaire asks participants to report on a 4-point scale (1=Strongly disagree - 4=Strongly agree) how much they agree with several statements about communicating with their child about sex (e.g., It would embarrass me to talk about sex and birth control with my child). Item responses will be averaged, and lower values represent a better outcome.
Time Frame: 1) pretest questionnaire; 2) posttest questionnaire - 4 weeks after pretest
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Resource 1 | Resource 2
Number analyzed (Participants) | 136 | 147
score on a scale | 1.62 (.0303) | 1.61 (.0297)
Statistical Analysis 1: Comparison: Resource 1 vs Resource 2; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = .87, Regression, Linear

8. Secondary Outcome: Change in Parent Outcome Expectancies Related to Communicating With Their Child About Relationship and Sexual Health From Pretest to Posttest
Description: Parent questionnaire asks participants to report on a 4-point scale (1=Strongly disagree - 4=Strongly agree) how much they agree with several statements about the outcomes of communicating with their child about sex (e.g., I will feel proud). Item responses will be averaged, and higher values represent a better outcome.
Time Frame: 1) pretest questionnaire; 2) posttest questionnaire - 4 weeks after pretest
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Resource 1 | Resource 2
Number analyzed (Participants) | 138 | 150
score on a scale | 3.11 (.0238) | 3.10 (.0235)
Statistical Analysis 1: Comparison: Resource 1 vs Resource 2; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = .8, Regression, Linear

9. Secondary Outcome: Change in Parent Self-efficacy to Engage in Communication With Their Child About Relationship and Sexual Health From Pretest to Posttest
Description: Parent questionnaire asks participants to report on a 7-point scale (1=not sure at all - 7=completely sure) how sure they are that they can explain to their child about several relationship and sexual health topics (e.g., how pregnancy happens). Item responses will be averaged, and higher values represent a better outcome.
Time Frame: 1) pretest questionnaire; 2) posttest questionnaire - 4 weeks after pretest
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Resource 1 | Resource 2
Number analyzed (Participants) | 138 | 150
score on a scale | 6.27 (.0652) | 6.20 (.063)
Statistical Analysis 1: Comparison: Resource 1 vs Resource 2; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = .32, Regression, Linear

10. Secondary Outcome: Change in Parent Reported Parent-child Communication Quality From Pretest to Posttest
Description: Parent questionnaire asks participants on a 4-point scale (1=Strongly disagree - 4=Strongly agree) how much they agree with several statements related to parent-child communication (e.g., My child and I can talk about almost anything.) Item responses will be averaged, and higher values represent a better outcome.
Time Frame: 1) pretest questionnaire; 2) posttest questionnaire - 4 weeks after pretest
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Resource 1 | Resource 2
Number analyzed (Participants) | 140 | 153
score on a scale | 3.14 (.0238) | 3.08 (.0233)
Statistical Analysis 1: Comparison: Resource 1 vs Resource 2; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = .03, Regression, Linear

11. Secondary Outcome: Change in Child Reported Parent-child Communication Quality From Pretest to Posttest
Description: Child questionnaire asks participants on a 4-point scale (1=Strongly disagree - 4=Strongly agree) how much they agree with several statements related to parent-child communication (e.g., My parent and I can talk about almost anything.) Item responses will be averaged, and higher values represent a better outcome.
Time Frame: 1) pretest questionnaire; 2) posttest questionnaire - 4 weeks after pretest
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Resource 1 | Resource 2
Number analyzed (Participants) | 128 | 145
score on a scale | 3.22 (.0387) | 3.13 (.0382)
Statistical Analysis 1: Comparison: Resource 1 vs Resource 2; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = .05, Regression, Linear

12. Secondary Outcome: Change in Parent Skepticism of Media Messages From Pretest to Posttest
Description: Parent questionnaire asks participants on a 4-point scale (1=Strongly disagree - 4=Strongly agree) how much they agree with several statements about media. Item responses will be averaged, and higher values represent a better outcome.
Time Frame: 1) pretest questionnaire; 2) posttest questionnaire - 4 weeks after pretest
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Resource 1 | Resource 2
Number analyzed (Participants) | 127 | 139
score on a scale | 3.41 (.0511) | 3.29 (.0501)
Statistical Analysis 1: Comparison: Resource 1 vs Resource 2; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = .04, Regression, Linear

13. Secondary Outcome: Change in Child Skepticism of Media Messages From Pretest to Posttest
Description: Child questionnaire asks participants on a 4-point scale (1=Strongly disagree - 4=Strongly agree) how much they agree with several statements about media. Item responses will be averaged, and higher values represent a better outcome.
Time Frame: 1) pretest questionnaire; 2) posttest questionnaire - 4 weeks after pretest
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Resource 1 | Resource 2
Number analyzed (Participants) | 119 | 125
score on a scale | 2.98 (.0527) | 2.94 (.0544)
Statistical Analysis 1: Comparison: Resource 1 vs Resource 2; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = .42, Regression, Linear

14. Secondary Outcome: Change in Parent Perceived Realism of Media Messages From Pretest to Posttest
Description: Parent questionnaire asks participants on a 4-point scale (1=Strongly disagree - 4=Strongly agree) how much they agree with several statements about media. Item responses will be averaged, and lower values represent a better outcome.
Time Frame: 1) pretest questionnaire; 2) posttest questionnaire - 4 weeks after pretest
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Resource 1 | Resource 2
Number analyzed (Participants) | 139 | 150
score on a scale | 2.00 (.0504) | 2.09 (.0494)
Statistical Analysis 1: Comparison: Resource 1 vs Resource 2; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = .11, Regression, Linear

15. Secondary Outcome: Change in Child Perceived Realism of Media Messages From Pretest to Posttest
Description: Child questionnaire asks participants on a 4-point scale (1=Strongly disagree - 4=Strongly agree) how much they agree with several statements about media. Item responses will be averaged, and lower values represent a better outcome.
Time Frame: 1) pretest questionnaire; 2) posttest questionnaire - 4 weeks after pretest
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Resource 1 | Resource 2
Number analyzed (Participants) | 129 | 142
score on a scale | 2.07 (.0567) | 2.3 (.0563)
Statistical Analysis 1: Comparison: Resource 1 vs Resource 2; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = .0003, Regression, Linear

16. Secondary Outcome: Change in Child Sexual Media Exposure From Pretest to Posttest
Description: Child questionnaire asks participants to report on a 4-point scale (1=Never - 4=Often) how frequently they consume various media (e.g., Think about your average week. How often do you watch television shows?), and the sexual content of the media they consume (e.g., How would you rate the amount of sexual content in the television shows you watch? No sexual content, A little sexual content, Some sexual content, A lot of sexual content). Lower values represent a better outcome.
Time Frame: 1) pretest questionnaire; 2) posttest questionnaire - 4 weeks after pretest
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Resource 1 | Resource 2
Number analyzed (Participants) | 122 | 134
score on a scale | 1.79 (.0434) | 1.79 (.0424)
Statistical Analysis 1: Comparison: Resource 1 vs Resource 2; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = .97, Regression, Linear

17. Secondary Outcome: Change in Child Risky Online Behaviors From Pretest to Posttest
Description: Child questionnaire asks participants to indicate on a 5-point scale (1=Never; 2=Rarely; 3=Sometimes; 4=Often; 5=Always) how often they have experienced several online situations (e.g., been exposed to sexual content online). Item responses will be averaged, and lower values represent a better outcome.
Time Frame: 1) pretest questionnaire; 2) posttest questionnaire - 4 weeks after pretest
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Resource 1 | Resource 2
Number analyzed (Participants) | 128 | 142
score on a scale | 1.43 (.0335) | 1.50 (.0327)
Statistical Analysis 1: Comparison: Resource 1 vs Resource 2; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = .08, Regression, Linear

18. Secondary Outcome: Change in Child Intentions to Engage in Sexual Activity From Pretest to Posttest
Description: The child questionnaire asks participants to report on a 4-point scale how likely it is that they will engage in sexual activity (e.g., How likely is it that you will have sex in the next year?) (1=Not likely at all, 2=Unlikely, 3=Likely, 4=Very likely) Participant's responses will be averaged, and lower values represent a better outcome.
Time Frame: 1) pretest questionnaire; 2) posttest questionnaire - 4 weeks after pretest
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Resource 1 | Resource 2
Number analyzed (Participants) | 129 | 141
score on a scale | 1.3891 (.0003) | 1.3892 (.0003)
Statistical Analysis 1: Comparison: Resource 1 vs Resource 2; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = .70, Regression, Linear

19. Secondary Outcome: Change in Willingness to Engage in Unwanted Sexual Activity From Pretest to Posttest
Description: The child questionnaire asks participants to report on a 4-point scale (1=Very unwilling - 4=Very willing) their willingness to engage in sexual activity if they were not sure that they wanted to. Lower values represent a better outcome.
Time Frame: 1) pretest questionnaire; 2) posttest questionnaire - 4 weeks after pretest
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Resource 1 | Resource 2
Number analyzed (Participants) | 128 | 140
score on a scale | 1.69 (.0579) | 1.83 (.0578)
Statistical Analysis 1: Comparison: Resource 1 vs Resource 2; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = .03, Regression, Linear

20. Secondary Outcome: Change in Parent Report of Parental Evaluative Media Mediation From Pretest to Posttest
Description: Parent questionnaire asks participants to rate on a 4-point scale (1=Never - 4=Often) how frequently the parent engages in evaluative media mediation related to media use and rules. Item responses will be averaged, and higher values represent a better outcome.
Time Frame: 1) pretest questionnaire; 2) posttest questionnaire - 4 weeks after pretest
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Resource 1 | Resource 2
Number analyzed (Participants) | 139 | 150
score on a scale | 3.21 (.0519) | 3.28 (.0518)
Statistical Analysis 1: Comparison: Resource 1 vs Resource 2; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = .29, Regression, Linear

21. Secondary Outcome: Change in Child Report of Parental Evaluative Media Mediation From Pretest to Posttest
Description: Child questionnaire asks participants to rate on a 4-point scale (1=Never - 4=Often) how frequently the parent engages in several evaluative mediation behaviors related to media use and rules.Item responses will be averaged, and higher values represent a better outcome.
Time Frame: 1) pretest questionnaire; 2) posttest questionnaire - 4 weeks after pretest; 3) follow-up questionnaire - 24 weeks after pretest
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Resource 1 | Resource 2
Number analyzed (Participants) | 128 | 143
score on a scale | 2.72 (.0688) | 2.79 (.0679)
Statistical Analysis 1: Comparison: Resource 1 vs Resource 2; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = .36, Regression, Linear

22. Secondary Outcome: Change in Child Attitudes About Teen Sex From Pretest to Posttest
Description: Child questionnaire asks participants to indicate on a 4-point scale (1=strongly disagree - 4=Strongly agree) how much they agree with several statements about teen sex. Item responses will be averaged, and lower values represent a better outcome.
Time Frame: 1) pretest questionnaire; 2) posttest questionnaire - 4 weeks after pretest
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Resource 1 | Resource 2
Number analyzed (Participants) | 128 | 143
score on a scale | 2.06 (.0433) | 2.08 (.0428)
Statistical Analysis 1: Comparison: Resource 1 vs Resource 2; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = .61, Regression, Linear

23. Secondary Outcome: Change in Sexual Abstinence Self-efficacy Form Pretest to Posttest
Description: Child questionnaire asks participants to indicate on a 4-point scale (1=Strongly disagree - 4=Strongly agree) how much they agree with several statements related to abstaining from sexual activity. Item responses will be averaged, and higher values represent a better outcome.
Time Frame: 1) pretest questionnaire; 2) posttest questionnaire - 4 weeks after pretest
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Resource 1 | Resource 2
Number analyzed (Participants) | 126 | 139
score on a scale | 3.5 (.0466) | 3.48 (.0465)
Statistical Analysis 1: Comparison: Resource 1 vs Resource 2; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = .72, Regression, Linear

24. Secondary Outcome: Change in Contraception Self-efficacy From Pretest to Posttest
Description: Child questionnaire asks participants to indicate on a 4-point scale (1=Strongly disagree - 4=Strongly agree) how much they agree with several statements related to contraception. Item responses will be averaged, and higher values represent a better outcome.
Time Frame: 1) pretest questionnaire; 2) posttest questionnaire - 4 weeks after pretest
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Resource 1 | Resource 2
Number analyzed (Participants) | 125 | 136
score on a scale | 2.97 (.07) | 2.82 (.0713)
Statistical Analysis 1: Comparison: Resource 1 vs Resource 2; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = .05, Regression, Linear

25. Secondary Outcome: Change in Supportive Parenting - Child Report From Pretest to Posttest
Description: Child questionnaire asks participants to indicate on a 4-point scale (1=Never - 4=Always) how much they agree with several statements related to how often their parent engages in certain behaviors (e.g., How often does your parent let you know they care about you?). Item responses will be averaged, and higher values represent a better outcome.
Time Frame: 1) pretest questionnaire; 2) posttest questionnaire - 4 weeks after pretest
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Resource 1 | Resource 2
Number analyzed (Participants) | 121 | 135
score on a scale | 3.5 (.0467) | 3.42 (.0458)
Statistical Analysis 1: Comparison: Resource 1 vs Resource 2; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = .09, Regression, Linear

26. Secondary Outcome: Change in Supportive Parenting - Parent Report From Pretest to Posttest
Description: Parent questionnaire asks participants to indicate on a 4-point scale (1=Never - 4=Always) how much they agree with several statements related to how often they engage in certain behaviors (e.g., How often do you let your child know you care about them?). Item responses will be averaged, and higher values represent a better outcome.
Time Frame: 1) pretest questionnaire; 2) posttest questionnaire - 4 weeks after pretest;
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Resource 1 | Resource 2
Number analyzed (Participants) | 141 | 152
score on a scale | 3.63 (.1329) | 3.62 (.0323)
Statistical Analysis 1: Comparison: Resource 1 vs Resource 2; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = .69, Regression, Linear

27. Secondary Outcome: Change in Parents Perceived Role in Child's Sexual Health Education From Pretest to Posttest
Description: The parent questionnaire asks, "I feel that someone else would do a better job teaching my child about sex and relationships." Parents respond to this question on a 4-point scale [Strongly disagree - Strongly agree]. Lower scores indicate more disagreement with the statement.
Time Frame: as for outcome 21
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Resource 1 | Resource 2
Number analyzed (Participants) | 135 | 146
score on a scale | 1.54 (.0526) | 1.64 (.0511)
Statistical Analysis 1: Comparison: Resource 1 vs Resource 2; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = .11, Regression, Linear

28. Secondary Outcome: Change in Frequency of Parent-child Sexual Health Discussions - Parent Report From Pretest to Posttest
Description: Parent questionnaires ask participants how frequently they engage in parent-child communication about sex and romantic relationships (1. Never; 2. Rarely; 3. Sometimes; 4. Often). Higher numbers represent a better outcome.
Time Frame: 1) pretest questionnaire; 2) posttest questionnaire - 4 weeks after pretest
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: score on a scale
Arm/Group | Resource 1 | Resource 2
Number analyzed (Participants) | 138 | 151
score on a scale | 2.89 (.0598) | 2.82 (.0584)
Statistical Analysis 1: Comparison: Resource 1 vs Resource 2; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = .27, Regression, Linear

29. Secondary Outcome: Change in Frequency of Parent-child Sexual Health Discussions - Child Report From Pretest to Posttest
Description: Child questionnaires ask participants how frequently they engage in parent-child communication about sex and relationships. (1. Never; 2. Rarely; 3. Sometimes; 4. Often). Higher numbers represent a better outcome.
Time Frame: 1) pretest questionnaire; 2) posttest questionnaire - 4 weeks after pretest
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Resource 1 | Resource 2
Number analyzed (Participants) | 136 | 145
score on a scale | 2.54 (.0613) | 2.57 (.0606)
Statistical Analysis 1: Comparison: Resource 1 vs Resource 2; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = .83, Regression, Linear

30. Secondary Outcome: Change in Perceived Media Message Completeness - Parent Report From Pretest to Posttest
Description: Participant views a print advertisement and parent questionnaire asks, "How complete is the information in this advertisement?" Participants respond to this question on a 5-point scale [Incomplete-Complete]. Lower scores represent a better outcome.
Time Frame: as for outcome 21
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Resource 1 | Resource 2
Number analyzed (Participants) | 140 | 151
score on a scale | 1.78 (.117) | 2.35 (.114)
Statistical Analysis 1: Comparison: Resource 1 vs Resource 2; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = .0001, Regression, Linear

31. Secondary Outcome: Change in Perceived Media Message Completeness - Child Report From Pretest to Posttest
Description: Participant views a print advertisement and child questionnaire asks, "How complete is the information in this advertisement?" Participants respond to this question on a 5-point scale [Incomplete-Complete]. Lower scores represent a better outcome.
Time Frame: 1) pretest questionnaire; 2) posttest questionnaire - 4 weeks after pretest
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Resource 1 | Resource 2
Number analyzed (Participants) | 123 | 134
score on a scale | 2.34 (.13) | 2.53 (.133)
Statistical Analysis 1: Comparison: Resource 1 vs Resource 2; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = .20, Regression, Linear

32. Secondary Outcome: Change in Parent Report of Parental Restrictive Media Mediation From Pretest to Posttest
Description: Parent questionnaire asks participants to rate on a 4-point scale (1=Never - 4=Often) how frequently the parent engages in several restrictive mediation behaviors related to media use and rules. Item responses will be averaged, and higher values represent a better outcome.
Time Frame: as for outcome 21
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Resource 1 | Resource 2
Number analyzed (Participants) | 139 | 150
score on a scale | 3.28 (.0545) | 3.17 (.0542)
Statistical Analysis 1: Comparison: Resource 1 vs Resource 2; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = .09, Regression, Linear

33. Secondary Outcome: Change in Child Report of Parental Restrictive Media Mediation From Pretest to Posttest
Description: Child questionnaire asks participants to rate on a 4-point scale (1=Never - 4=Often) how frequently the parent engages in several restrictive mediation behaviors related to media use and rules. Item responses will be averaged, and higher values represent a better outcome.
Time Frame: 1) pretest questionnaire; 2) posttest questionnaire - 4 weeks after pretest
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Resource 1 | Resource 2
Number analyzed (Participants) | 128 | 143
score on a scale | 2.66 (.0737) | 2.7 (.0725)
Statistical Analysis 1: Comparison: Resource 1 vs Resource 2; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = .62, Regression, Linear

34. Secondary Outcome: Change in Willingness to Engage in Unprotected Sexual Activity From Pretest to Posttest
Description: The child questionnaire asks participants to report on a 4-point scale (1=Very unwilling - 4=Very willing) their willingness to engage in unprotected sexual activity. Lower values represent a better outcome.
Time Frame: 1) pretest questionnaire; 2) posttest questionnaire - 4 weeks after pretest
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Resource 1 | Resource 2
Number analyzed (Participants) | 125 | 131
score on a scale | 1.34376 (.0001) | 1.34378 (.0001)
Statistical Analysis 1: Comparison: Resource 1 vs Resource 2; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = .29, Regression, Linear

35. Secondary Outcome: Change in Attitudes Toward Teen Contraception Use - Child Report From Pretest to Posttest
Description: Child questionnaire asks participant to indicate their extent of agreement or disagreement on a 4-point scale [strongly disagree - strongly agree] with several statements about teen contraception us (e.g., condoms should always be used if a teen has sex.) Higher score indicates more favorable outcome.
Time Frame: 1) pretest questionnaire; 2) posttest questionnaire - 4 weeks after pretest
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Resource 1 | Resource 2
Number analyzed (Participants) | 128 | 141
score on a scale | 3.53 (.0489) | 3.45 (.0485)
Statistical Analysis 1: Comparison: Resource 1 vs Resource 2; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = .14, Regression, Linear

36. Secondary Outcome: Change in Intentions to Communicate With a Medical Professional From Pretest to Posttest
Description: Child questionnaire asks participants to indicate "Before deciding to have sex, how likely would you be to talk to your doctor or other medical professional?" Participants indicate their likelihood on a 4-point scale [1=Not at all likely; 2=Unlikely; 3=Likely; 4=Very likely]. Higher score indicates a more favorable outcome.
Time Frame: 1) pretest questionnaire; 2) posttest questionnaire - 4 weeks after pretest
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Resource 1 | Resource 2
Number analyzed (Participants) | 124 | 130
score on a scale | 2.28 (.0916) | 1.99 (.0931)
Statistical Analysis 1: Comparison: Resource 1 vs Resource 2; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = .008, Regression, Linear

37. Secondary Outcome: Change in Attitudes Toward Sexual Communication - Child Report From Pretest to Posttest
Description: Child questionnaire asks participants to indicate their level of agreement on a 4-point scale [Strongly disagree - Strongly agree] to several statements about sexual communication (e.g., Before deciding to have sex, I believe teens should talk with their partner about pregnancy.). Higher scores indicate more favorable outcome.
Time Frame: 1) pretest questionnaire; 2) posttest questionnaire - 4 weeks after pretest
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Resource 1 | Resource 2
Number analyzed (Participants) | 126 | 141
score on a scale | 3.42 (.0506) | 3.29 (.0501)
Statistical Analysis 1: Comparison: Resource 1 vs Resource 2; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = .02, Regression, Linear

38. Secondary Outcome: Change in Perceived Parental Permissiveness Toward Teen Sex - Child Report From Pretest to Posttest
Description: Youth reported on their perceptions of their parent's permissiveness regarding their sexual activity (five items; 4-point Likert scale; Strongly disagree to Strongly agree; α=.76). Sample items include "My parent would approve of my having sex at this time in my life." Higher values indicate that the youth believes their parent is more permissive of their sexual activity as a teen.
Time Frame: 1) pretest questionnaire; 2) posttest questionnaire - 4 weeks after pretest
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Resource 1 | Resource 2
Number analyzed (Participants) | 121 | 138
score on a scale | 1.44 (.0489) | 1.56 (.0477)
Statistical Analysis 1: Comparison: Resource 1 vs Resource 2; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = .03, Regression, Linear

39. Secondary Outcome: Change in Normative Beliefs About Teen Sex - Child Report From Pretest to Posttest
Description: Youth reported on the proportion of teens they believe are engaging in sexual behavior: "What percentage of teens are having sex? [(0% (no teens) to 100% (all teens)]."
Time Frame: as for outcome 21
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Resource 1 | Resource 2
Number analyzed (Participants) | 121 | 138
score on a scale | 48.3 (2.59) | 49.4 (2.35)
Statistical Analysis 1: Comparison: Resource 1 vs Resource 2; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = .69, Regression, Linear

40. Secondary Outcome: Change in Family Having Rules About Media Use - Parent Report From Pretest to Posttest
Description: Parent questionnaire asked parents to report about the media rules in their family, "Does your family have rules about media use? (one item; Yes, No, Unsure).
Time Frame: 1) pretest questionnaire; 2) posttest questionnaire - 4 weeks after pretest
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Resource 1 | Resource 2
Number analyzed (Participants) | 126 | 144
score on a scale | 1.48 (.0001) | 1.48 (.0001)
Statistical Analysis 1: Comparison: Resource 1 vs Resource 2; Test type: Equivalence — Binary outcomes were assessed with logistic regression; p = .4, Regression, Logistic

41. Secondary Outcome: Change in Awareness of Family Having Rules About Media Use - Child Report From Pretest to Posttest
Description: Child questionnaire asked child to report about the media rules in their family, "Does your family have rules about media use? (one item; Yes, No, Unsure). Participants selected either 'Yes,' 'No,' or 'Unsure' (no and unsure were combined for analyses).
Time Frame: 1) pretest questionnaire; 2) posttest questionnaire - 4 weeks after pretest
Population: as for outcome 1
Measure: Number; unit: odds ratio
Arm/Group | Resource 1 | Resource 2
Number analyzed (Participants) | 126 | 144
odds ratio | 1.169 | .311
Statistical Analysis 1: Comparison: Resource 1 vs Resource 2; Test type: Equivalence — Binary outcomes were assessed with logistic regression; p = .02, Regression, Logistic

42. Secondary Outcome: Change in Parental Perceived Importance of Parent-child Communication About Relationship and Sexual Health From Pretest to Follow-up
Description: as for outcome 5
Time Frame: 1) pretest questionnaire; 2) follow-up questionnaire - 24 weeks after pretest
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Resource 1 | Resource 2
Number analyzed (Participants) | 147 | 141
score on a scale | 3.69 (.03) | 3.66 (.03)
Statistical Analysis 1: Comparison: Resource 1 vs Resource 2; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; p = .27, Regression, Linear

43. Secondary Outcome: Change in Parent Level of Comfort With Parent-child Communication About Relationship and Sexual Health From Pretest to Follow-up
Description: as for outcome 6
Time Frame: 1) pretest questionnaire; 2) follow-up questionnaire - 24 weeks after pretest
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Resource 1 | Resource 2
Number analyzed (Participants) | 148 | 143
score on a scale | 3.48 (.05) | 3.52 (.04)
Statistical Analysis 1: Comparison: Resource 1 vs Resource 2; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; p = .31, Regression, Linear

44. Secondary Outcome: Change in Parent Reservations About Parent-child Communication About Relationship and Sexual Health From Pretest to Follow-up
Description: as for outcome 7
Time Frame: 1) pretest questionnaire; 2) follow-up questionnaire - 24 weeks after pretest
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Resource 1 | Resource 2
Number analyzed (Participants) | 144 | 139
score on a scale | 1.63 (.05) | 1.57 (.05)
Statistical Analysis 1: Comparison: Resource 1 vs Resource 2; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; p = .11, Regression, Linear

45. Secondary Outcome: Change in Parent Outcome Expectancies Related to Communicating With Their Child About Relationship and Sexual Health From Pretest to Follow-up
Description: as for outcome 8
Time Frame: 1) pretest questionnaire; 2) follow-up questionnaire - 24 weeks after pretest
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Resource 1 | Resource 2
Number analyzed (Participants) | 146 | 142
score on a scale | 3.09 (.03) | 3.08 (.03)
Statistical Analysis 1: Comparison: Resource 1 vs Resource 2; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; p = .89, Regression, Linear

46. Secondary Outcome: Change in Parent Self-efficacy to Engage in Communication With Their Child About Relationship and Sexual Health From Pretest to Follow-up
Description: as for outcome 9
Time Frame: 1) pretest questionnaire; 2) follow-up questionnaire - 24 weeks after pretest
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Resource 1 | Resource 2
Number analyzed (Participants) | 147 | 142
score on a scale | 6.27 (.08) | 6.33 (.08)
Statistical Analysis 1: Comparison: Resource 1 vs Resource 2; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; p = .41, Regression, Linear

47. Secondary Outcome: Change in Parent Reported Parent-child Communication Quality From Pretest to Follow-up
Description: as for outcome 10
Time Frame: 1) pretest questionnaire; 2) follow-up questionnaire - 24 weeks after pretest
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Resource 1 | Resource 2
Number analyzed (Participants) | 146 | 140
score on a scale | 2.92 (.04) | 2.92 (.04)
Statistical Analysis 1: Comparison: Resource 1 vs Resource 2; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; p = .93, Regression, Linear

48. Secondary Outcome: Change in Child Reported Parent-child Communication Quality From Pretest to Follow-up
Description: as for outcome 11
Time Frame: 1) pretest questionnaire; 2) follow-up questionnaire - 24 weeks after pretest
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Resource 1 | Resource 2
Number analyzed (Participants) | 138 | 143
score on a scale | 3.18 (.04) | 3.17 (.04)
Statistical Analysis 1: Comparison: Resource 1 vs Resource 2; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; p = .83, Regression, Linear

49. Secondary Outcome: Change in Parent Skepticism of Media Messages From Pretest to Follow-up
Description: as for outcome 12
Time Frame: 1) pretest questionnaire; 2) follow-up questionnaire - 24 weeks after pretest
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Resource 1 | Resource 2
Number analyzed (Participants) | 130 | 125
score on a scale | 3.38 (.07) | 3.26 (.07)
Statistical Analysis 1: Comparison: Resource 1 vs Resource 2; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; p = .04, Regression, Linear

50. Secondary Outcome: Change in Child Skepticism of Media Messages From Pretest to Follow-up
Description: as for outcome 13
Time Frame: 1) pretest questionnaire; 2) follow-up questionnaire - 24 weeks after pretest
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Resource 1 | Resource 2
Number analyzed (Participants) | 113 | 120
score on a scale | 3.03 (.07) | 2.93 (.07)
Statistical Analysis 1: Comparison: Resource 1 vs Resource 2; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; p = .13, Regression, Linear

51. Secondary Outcome: Change in Child Perceived Realism of Media Messages From Pretest to Follow-up
Description: as for outcome 15
Time Frame: 1) pretest questionnaire; 2) follow-up questionnaire - 24 weeks after pretest
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Resource 1 | Resource 2
Number analyzed (Participants) | 139 | 143
score on a scale | 2.3 (.08) | 2.34 (.08)
Statistical Analysis 1: Comparison: Resource 1 vs Resource 2; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; p = .56, Regression, Linear

52. Secondary Outcome: Change in Child Sexual Media Exposure From Pretest to Follow-up
Description: as for outcome 16
Time Frame: 1) pretest questionnaire; 2) follow-up questionnaire - 24 weeks after pretest
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Resource 1 | Resource 2
Number analyzed (Participants) | 123 | 126
score on a scale | 17.6 (1.46) | 17.5 (1.51)
Statistical Analysis 1: Comparison: Resource 1 vs Resource 2; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; p = .96, Regression, Linear

53. Secondary Outcome: Change in Child Risky Online Behaviors From Pretest to Follow-up
Description: as for outcome 17
Time Frame: 1) pretest questionnaire; 2) follow-up questionnaire - 24 weeks after pretest
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Resource 1 | Resource 2
Number analyzed (Participants) | 138 | 143
score on a scale | 1.51 (.06) | 1.56 (.05)
Statistical Analysis 1: Comparison: Resource 1 vs Resource 2; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; p = .35, Regression, Linear

54. Secondary Outcome: Change in Child Intentions to Engage in Sexual Activity From Pretest to Follow-up
Description: as for outcome 18
Time Frame: 1) pretest questionnaire; 2) follow-up questionnaire - 24 weeks after pretest
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Resource 1 | Resource 2
Number analyzed (Participants) | 138 | 140
score on a scale | 1.61 (.09) | 1.52 (.09)
Statistical Analysis 1: Comparison: Resource 1 vs Resource 2; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; p = .24, Regression, Linear

55. Secondary Outcome: Change in Willingness to Engage in Unwanted Sexual Activity From Pretest to Follow-up
Description: as for outcome 19
Time Frame: 1) pretest questionnaire; 2) follow-up questionnaire - 24 weeks after pretest
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Resource 1 | Resource 2
Number analyzed (Participants) | 137 | 140
score on a scale | 1.93 (.09) | 1.83 (.09)
Statistical Analysis 1: Comparison: Resource 1 vs Resource 2; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; p = .2, Regression, Linear

56. Secondary Outcome: Change in Parent Report of Parental Evaluative Media Mediation From Pretest to Follow-up
Description: as for outcome 20
Time Frame: 1) pretest questionnaire; 2) follow-up questionnaire - 24 weeks after pretest
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Resource 1 | Resource 2
Number analyzed (Participants) | 145 | 142
score on a scale | 3.13 (.07) | 3.22 (.06)
Statistical Analysis 1: Comparison: Resource 1 vs Resource 2; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; p = .18, Regression, Linear

57. Secondary Outcome: Change in Child Report of Parental Evaluative Media Mediation From Pretest to Follow-up
Description: as for outcome 21
Time Frame: 1) pretest questionnaire; 3) follow-up questionnaire - 24 weeks after pretest
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Resource 1 | Resource 2
Number analyzed (Participants) | 139 | 143
score on a scale | 2.75 (.09) | 2.78 (.09)
Statistical Analysis 1: Comparison: Resource 1 vs Resource 2; To examine intervention effects, a residual difference score approach was used to provide an estimate of change from baseline and is assessed by regressing follow-up scores onto baseline scores and the treatment variables; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; p = .67, Regression, Linear

58. Secondary Outcome: Change in Child Attitudes About Teen Sex From Pretest to Follow-up
Description: as for outcome 22
Time Frame: 1) pretest questionnaire; 2) follow-up questionnaire - 24 weeks after pretest
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Resource 1 | Resource 2
Number analyzed (Participants) | 139 | 143
score on a scale | 2.1 (.06) | 2.13 (.06)
Statistical Analysis 1: Comparison: Resource 1 vs Resource 2; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; p = .57, Regression, Linear

59. Secondary Outcome: Change in Sexual Abstinence Self-efficacy From Pretest to Follow-up
Description: as for outcome 23
Time Frame: 1) pretest questionnaire; 2) follow-up questionnaire - 24 weeks after pretest
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Resource 1 | Resource 2
Number analyzed (Participants) | 138 | 139
score on a scale | 3.38 (.07) | 3.4 (.07)
Statistical Analysis 1: Comparison: Resource 1 vs Resource 2; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; p = .65, Regression, Linear

60. Secondary Outcome: Change in Contraception Self-efficacy From Pretest to Follow-up
Description: as for outcome 24
Time Frame: 1) pretest questionnaire; 2) follow-up questionnaire - 24 weeks after pretest
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Resource 1 | Resource 2
Number analyzed (Participants) | 136 | 135
score on a scale | 3.09 (.12) | 3.03 (.12)
Statistical Analysis 1: Comparison: Resource 1 vs Resource 2; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; p = .84, Regression, Linear

61. Secondary Outcome: Change in Supportive Parenting - Child Report From Pretest to Follow-up
Description: as for outcome 25
Time Frame: 1) pretest questionnaire; 2) follow-up questionnaire - 24 weeks after pretest
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Resource 1 | Resource 2
Number analyzed (Participants) | 134 | 133
score on a scale | 3.63 (.07) | 3.48 (.07)
Statistical Analysis 1: Comparison: Resource 1 vs Resource 2; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; p = .02, Regression, Linear

62. Secondary Outcome: Change in Supportive Parenting - Parent Report Form Pretest to Follow-up
Description: as for outcome 26
Time Frame: 1) pretest questionnaire; 2) follow-up questionnaire - 24 weeks after pretest
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Resource 1 | Resource 2
Number analyzed (Participants) | 147 | 143
score on a scale | 3.63 (.04) | 3.64 (.04)
Statistical Analysis 1: Comparison: Resource 1 vs Resource 2; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; p = .65, Regression, Linear

63. Secondary Outcome: Change in Parents Perceived Role in Child's Sexual Health Education From Pretest to Follow-up
Description: as for outcome 27
Time Frame: 1) pretest questionnaire; 2) follow-up questionnaire - 24 weeks after pretest
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Resource 1 | Resource 2
Number analyzed (Participants) | 140 | 136
score on a scale | 1.60 (.09) | 1.46 (.09)
Statistical Analysis 1: Comparison: Resource 1 vs Resource 2; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; p = .09, Regression, Linear

64. Secondary Outcome: Change in Frequency of Parent-child Sexual Health Discussions - Parent Report From Pretest to Follow-up
Description: as for outcome 28
Time Frame: 1) pretest questionnaire; 3) follow-up questionnaire - 24 weeks after pretest
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: score on a scale
Arm/Group | Resource 1 | Resource 2
Number analyzed (Participants) | 147 | 140
score on a scale | 2.94 (.08) | 2.94 (.08)
Statistical Analysis 1: Comparison: Resource 1 vs Resource 2; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; p = .95, Regression, Linear

65. Secondary Outcome: Change in Frequency of Parent-child Sexual Health Discussions - Child Report From Pretest to Follow-up
Description: as for outcome 29
Time Frame: 1) pretest questionnaire; 2) ) follow-up questionnaire - 24 weeks after pretest
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Resource 1 | Resource 2
Number analyzed (Participants) | 136 | 141
score on a scale | 2.70 (.09) | 2.68 (.09)
Statistical Analysis 1: Comparison: Resource 1 vs Resource 2; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; p = .47, Regression, Linear

66. Secondary Outcome: Change in Perceived Media Message Completeness - Parent Report From Pretest to Follow-up
Description: as for outcome 30
Time Frame: 1) pretest questionnaire; 2) follow-up questionnaire - 24 weeks after pretest
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Resource 1 | Resource 2
Number analyzed (Participants) | 146 | 141
score on a scale | 1.85 (.16) | 2.31 (.16)
Statistical Analysis 1: Comparison: Resource 1 vs Resource 2; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; p = .003, Regression, Linear

67. Secondary Outcome: Change in Perceived Media Message Completeness - Child Report From Pretest to Follow-up
Description: as for outcome 31
Time Frame: 1) pretest questionnaire; 2) follow-up questionnaire - 24 weeks after pretest
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Resource 1 | Resource 2
Number analyzed (Participants) | 134 | 137
score on a scale | 2.5 (.18) | 2.54 (.18)
Statistical Analysis 1: Comparison: Resource 1 vs Resource 2; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; p = .77, Regression, Linear

68. Secondary Outcome: Change in Parent Report of Parental Restrictive Media Mediation From Pretest to Follow-up
Description: as for outcome 32
Time Frame: 1) pretest questionnaire; 2) follow-up questionnaire - 24 weeks after pretest
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Resource 1 | Resource 2
Number analyzed (Participants) | 145 | 142
score on a scale | 3.25 (.07) | 3.03 (.07)
Statistical Analysis 1: Comparison: Resource 1 vs Resource 2; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; p < .001, Regression, Linear

69. Secondary Outcome: Change in Child Report of Parental Restrictive Media Mediation From Pretest to Follow-up
Description: as for outcome 33
Time Frame: 1) pretest questionnaire; 2) follow-up questionnaire - 24 weeks after pretest
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Resource 1 | Resource 2
Number analyzed (Participants) | 139 | 143
score on a scale | 2.76 (.1) | 2.6 (.1)
Statistical Analysis 1: Comparison: Resource 1 vs Resource 2; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; p = .06, Regression, Linear

70. Secondary Outcome: Change in Willingness to Engage in Unprotected Sexual Activity From Pretest to Follow-up
Description: as for outcome 34
Time Frame: 1) pretest questionnaire; 2) follow-up questionnaire - 24 weeks after pretest
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Resource 1 | Resource 2
Number analyzed (Participants) | 134 | 131
score on a scale | 1.39 (.001) | 1.39 (.001)
Statistical Analysis 1: Comparison: Resource 1 vs Resource 2; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; p = .91, Regression, Linear

71. Secondary Outcome: Change in Attitudes Toward Teen Contraception Use - Child Report From Pretest to Follow-up
Description: as for outcome 35
Time Frame: 1) pretest questionnaire; 2) follow-up questionnaire - 24 weeks after pretest
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Resource 1 | Resource 2
Number analyzed (Participants) | 139 | 141
score on a scale | 3.37 (.07) | 3.38 (.07)
Statistical Analysis 1: Comparison: Resource 1 vs Resource 2; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; p = .95, Regression, Linear

72. Secondary Outcome: Change in Intentions to Communicate With a Medical Professional From Pretest to Follow-up
Description: as for outcome 36
Time Frame: 1) pretest questionnaire; 2) follow-up questionnaire - 24 weeks after pretest
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Resource 1 | Resource 2
Number analyzed (Participants) | 133 | 132
score on a scale | 2.3 (.14) | 2.12 (.13)
Statistical Analysis 1: Comparison: Resource 1 vs Resource 2; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; p = .12, Regression, Linear

73. Secondary Outcome: Change in Attitudes Toward Sexual Communication - Child Report From Pretest to Follow-up
Description: as for outcome 37
Time Frame: 1) pretest questionnaire; 2) follow-up questionnaire - 24 weeks after pretest
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Resource 1 | Resource 2
Number analyzed (Participants) | 138 | 141
score on a scale | 3.4 (.07) | 3.4 (.07)
Statistical Analysis 1: Comparison: Resource 1 vs Resource 2; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; p = .98, Regression, Linear

74. Secondary Outcome: Change in Perceived Parental Permissiveness Toward Teen Sex - Child Report From Pretest to Follow-up
Description: as for outcome 38
Time Frame: 1) pretest questionnaire; 2) follow-up questionnaire - 24 weeks after pretest
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Resource 1 | Resource 2
Number analyzed (Participants) | 124 | 126
score on a scale | 1.68 (.07) | 1.66 (.07)
Statistical Analysis 1: Comparison: Resource 1 vs Resource 2; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; p = .57, Regression, Linear

75. Secondary Outcome: Change in Normative Beliefs About Teen Sex - Child Report From Pretest to Follow-up
Description: as for outcome 39
Time Frame: 1) pretest questionnaire; 2) follow-up questionnaire - 24 weeks after pretest
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Resource 1 | Resource 2
Number analyzed (Participants) | 76 | 88
score on a scale | 50.4 (4.02) | 50.3 (3.91)
Statistical Analysis 1: Comparison: Resource 1 vs Resource 2; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; p = .98, Regression, Linear

76. Secondary Outcome: Change in Family Having Rules About Media Use - Parent Report From Pretest to Follow-up
Description: as for outcome 40
Time Frame: 1) pretest questionnaire;2) follow-up questionnaire - 24 weeks after pretest
Population: as for outcome 1
Measure: Number; unit: odds ratio
Arm/Group | Resource 1 | Resource 2
Number analyzed (Participants) | 148 | 142
odds ratio | 7.76 | 6.77
Statistical Analysis 1: Comparison: Resource 1 vs Resource 2; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; p = .07, Regression, Linear

77. Secondary Outcome: Change in Awareness of Family Having Rules About Media Use - Child Report From Pretest to Follow-up
Description: as for outcome 41
Time Frame: 1) pretest questionnaire; 2)follow-up questionnaire - 24 weeks after pretest
Population: as for outcome 1
Measure: Number; unit: odds ratio
Arm/Group | Resource 1 | Resource 2
Number analyzed (Participants) | 138 | 142
odds ratio | 1.11 | .35
Statistical Analysis 1: Comparison: Resource 1 vs Resource 2; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; p = .02, Regression, Linear

78. Secondary Outcome: Change in Parent Perceived Realism of Media Messages From Pretest to Follow-up
Description: as for outcome 14
Time Frame: 1) pretest questionnaire; 2) follow-up - 24 weeks after pretest
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Resource 1 | Resource 2
Number analyzed (Participants) | 144 | 138
score on a scale | 2.0 (.07) | 2.08 (.07)
Statistical Analysis 1: Comparison: Resource 1 vs Resource 2; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; p = .15, Regression, Linear

ADVERSE EVENTS:
Time Frame: Research staff members scanned the incoming online questionnaire data on a regularly basis and recorded any problems seen or concerns about any participants over the study timeframe (approx. 6 months).
Description: Study risks were defined as discomfort with assessment procedures/content, or breach of confidentiality. Measures were taken to provide confidentiality with respect to questionnaire responses and program process data.To minimize the risk of discomfort for participants, participants could skip any question and quit participation at any time. Research staff scanned the incoming data on a regularly basis to record any concerns about any participants. No adverse events were reported.
Arm/Group | Resource 1 | Resource 2
All-Cause Mortality (participants affected / at risk) | 0/358 | 0/372
Serious Adverse Events (participants affected / at risk) | 0/358 | 0/372
Other Adverse Events (participants affected / at risk) | 0/358 | 0/372

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-30): https://cdn.clinicaltrials.gov/large-docs/51/NCT03655951/Prot_SAP_000.pdf